CLINICAL TRIAL: NCT06030817
Title: A Prospective Study to Explore the Performance and Efficacy of 99mTc-CNDG Injection in Malignant Tumors
Brief Title: 99mTc-CNDG Injection in the Diagnosis of Malignant Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: K1999
Record Dates: First submitted 2023-09-03; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-08

CONDITIONS: Malignant Tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 99mTc-CNDG SPECT/CT (Experimental): Inject 99mTc-CNDG and then perform SPECT/CT scan.
  Interventions: Diagnostic Test: 99mTc-CNDG SPECT/CT

INTERVENTIONS:
Diagnostic Test: 99mTc-CNDG SPECT/CT — Explore the imaging characteristics of 99mTc-CNDG and its diagnostic efficacy in tumor patients.

SUMMARY:
Currently, 18F-fluorodeoxyglucose (18F-FDG) is the most widely used tumor imaging agent in clinical practice. However, the production of 18F requires accelerators and is associated with relatively high diagnostic costs, which to some extent limits its widespread clinical application. In comparison to Positron Emission Tomography (PET), Single Photon Emission Computed Tomography (SPECT) devices are more abundant and offer lower diagnostic expenses. With the utilization of Cadmium Zinc Telluride (CZT) crystals in SPECT and advancements in image reconstruction techniques, the resolution and sensitivity of SPECT is continually improving. Therefore, the development of a simplified and cost-effective novel SPECT tumor imaging agent holds significant practical significance. This study involved the design and synthesis of a glucose-derived ligand with a linker containing seven methylene units and an isonitrile group (CN7DG). The CN7DG ligand was labeled with 99mTc to prepare a more lipophilic 99mTc-CN7DG complex, aiming to investigate a novel SPECT imaging agent for tumor imaging.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old
* Patients diagnosed with malignant glioma, colorectal cancer, pancreatic cancer, lung cancer, breast cancer, or other malignant tumors through imaging techniques such as MRI, CT, and ultrasound, and who are scheduled for surgical resection or biopsy
* Solid tumor sizes greater than 2cm
* Voluntarily agree to participate and sign an informed consent form
* Can provide complete surgical records, pathological results, control data, and clinical follow-up results

Exclusion Criteria:

* Pre-treatment such as chemotherapy and targeted therapy has been administered
* Pregnancy and breastfeeding
* Claustrophobia
* The condition is severe and difficult to cooperate with
* Unable to obtain relevant control imaging data and clinical information

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-08-11 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Uptake value of 99mTc-CNDG in malignant tumors | through study completion, an average of 1 year
  The uptake value was measured in the malignant lesions on 99mTc-CNDG SPECT/CT.
Lesions detected by 99mTc-CNDG SPECT/CT | through study completion, an average of 1 year
  The number of target lesions was calculated by 99mTc-CNDG SPECT/CT
Compared with 18F-FDG PET/CT or CECT | through study completion, an average of 1 year
  The number of lesions detected by 99mTc-CNDG SPECT/CT was compared with 18F-FDG PET/CT or CECT

CONTACTS AND LOCATIONS:
Overall Officials: Hongli Jing, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China